CLINICAL TRIAL: NCT04266470
Title: Monitoring Blood Flow and Metabolic Activity in Malignant Tissue of Head and Neck Region Using the Lara Device
Brief Title: Monitoring Blood Flow and Metabolic Activity in Malignant Tissue of Head and Neck Region
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is no longer feasible at our site.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00056907; P30CA012197 (NIH); WFBCCC 01919 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Monitoring blood flow; Metabolic activity in malignant tissue - head/ neck; Tumor response to therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lara Device Scan (Experimental): This imaging study will be obtained strictly for the research purposes of mid-treatment assessment of blood flow and uptake kinetics analysis
  Interventions: Device: Lara Scan; Diagnostic Test: PET/CT Scan - Pre-treatment and Post-treatment

INTERVENTIONS:
Device: Lara Scan — Four (4) sensors will be placed prior to the injection of 18 F-fludeoxyglucose (18FDG) at the following sites: 7 cm above injection site; injection site; surface of palpable presumed malignant tissue; palpable carotid artery.
  Standard doses of 18-FDG will be injected per Department of Radiology protocols
  All injections will be evaluated to insure the total dose of 18-FDG has been injected. Injections resulting in moderate to severe extravasations, as interpreted by Lara software, will be segregated and evaluated on an individual basis.
  The sensors will remain in place for 60 minutes during the 18-FDG uptake period with the patient in a reclined chair.
  After the uptake time is complete, the sensors will be removed by the technologist and the participant will be released.
  The study team will then upload the sensor data to a personal computer in the treatment planning room where it will be coded and processed as a Lara scan.
Diagnostic Test: PET/CT Scan - Pre-treatment and Post-treatment — The PET/CT imaging will be conducted according to standard of care. The main alteration to process flow will be the addition of the Lucerno sensors just prior to the injection of the PET material.

SUMMARY:
This study will investigate the ability of Lucerno Dynamics Lara sensor when placed on the palpable carotid artery (or femoral artery) to monitor blood flow following the injection of 18-FDG and to distinguish peak flow in tumor versus tissue uptake. Investigators will then assess if differences in tumor versus tissue correlates with tumor response.

DETAILED DESCRIPTION:
Primary Objective: To determine if Lara sensors placed over the carotid and femoral arteries can measure the plasma activity of 18 F-fludeoxyglucose (18-FDG) at time of injection and determine if that peak activity in the artery can be distinguished from peak activity in malignant tissue to provide enough information to obtain the arterial input function.

Secondary Objective: To evaluate changes (baseline to post treatment) in tissue uptake at first pass (AUC and time to peak blood flow) and during the 60-minute period (metabolic activity) leading to the , positron emission tomography (PET) scan. This data is to be collected from the Lucerno Device placed over the carotid and femoral arteries monitoring 18 F-fludeoxyglucose (18-FDG) activity in blood and malignant tissue throughout the pre positron emission tomography (PET) scan period.

ELIGIBILITY:
Inclusion Criteria

* Squamous cell carcinoma of the nasopharynx, oral cavity, oropharynx or hypopharynx with palpable adenopathy in the neck. Biopsy proven within the last 90 days.
* Squamous cell carcinoma of the larynx regardless of lymph node status. Biopsy proven within the last 90 days.
* Age 18 or greater.
* Receiving definitive radiation therapy at Wake Forest University with or without concurrent systematic therapy.
* Participants must be able to provide study specific informed consent prior to study entry.
* Presence of metastatic disease is not an exclusion criteria provided subject will be receiving definitive doses of radiation to the local and regional disease.

Exclusion Criteria

* Cancers of the head and neck other than those stated above. This would include squamous cell carcinoma of unknown primary.
* No measurable disease in the head and neck (ie planned adjuvant radiation therapy for allowable cancers with high risk pathology following definitive surgery).
* Persons receiving less than curative doses of radiation.
* Age under 18
* Unable or unwilling to tolerate PET/CT scan
* Unable or unwilling to receive definitive treatment of their cancer at Wake Forest University
* Pregnant women
* Participants who present having already undergone a PET/CT will not be eligible for this study-because an important element of this trial is the assessment of 18-FDG uptake changes in response to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Tests That Input Function (IF) Could Be Calculated | At baseline
  If input function can be calculated on five (5) or more (out of 10) patients, then investigators will consider this a feasible procedure. Input function is calculated using time-activity curves (TAC) from the arterial blood flow detector and integrating the signal over time. Peak and minimum values of each of the four (4) Lara detector time-activity curves (TAC) will be recorded to determine a range of expected values and if they are different.

SECONDARY OUTCOMES:
Change in Areas Under the Curve (AUC) Measurements | Baseline up to 120 days after completion of treatment
  Investigators will use a repeated measures linear model with change in areas under the curve as the outcome and time from baseline and the baseline area under the curve as predictors. From the model investigators will report the estimated change at the post treatment Lara measurement. Participants should have three measurements of area under the curve (baseline, mid-treatment, 3-week measurement prior to PET scan).
Change in Time to Peak Arterial Blood Flow | Baseline up to 120 days after completion of treatment
  Investigators will use a repeated measures linear model with change in areas under the curve as the outcome and time from baseline and the baseline area under the curve as predictors. From the model investigators will report the estimated change at the post treatment Lara measurement. Participants should have three measurements of area under the curve (baseline, mid-treatment, 3-week measurement prior to PET scan).

OTHER OUTCOMES:
Tumor Response | Baseline and 120 days after completion of treatment
  A correlation will be calculated between areas under change and percent change in tumor size.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Frizzell, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No